CLINICAL TRIAL: NCT06215807
Title: Femtosecond Laser Arcuate Keratotomy Versus Toric Intraocular Lens Implantation in Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 82201158; 82201158 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Cataract; Astigmatism
Keywords: Astigmatism correction; Femtosecond laser arcuate keratotomy; Toric intraocular lens implantation; Femtosecond laser-assisted cataract surgery
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femtosecond laser arcuate keratotomy (Active Comparator): femtosecond laser arcuate keratotomy will be designed using Donnenfeld nomogram.
  Interventions: Procedure: Femtosecond laser arcuate keratotomy
- Toric intraocular lens implantation (Active Comparator): The Toric IOL power and alignment axis were calculated using the online calculator available at https://www.tecnistoriccalc.com
  Interventions: Procedure: Toric intraocular lens implantation

INTERVENTIONS:
Procedure: Femtosecond laser arcuate keratotomy — The patient will receive femtosecond laser arcuate keratotomy and femtosecond laser-assisted cataract surgery with implantation of a monofocal intraocular lens in one eye.
  Arms: Femtosecond laser arcuate keratotomy
Procedure: Toric intraocular lens implantation — The patient will receive femtosecond laser-assisted cataract surgery with implantation of a Toric monofocal intraocular lens in the contralateral eye.
  Arms: Toric intraocular lens implantation

SUMMARY:
In modern cataract surgery, residual astigmatism continues to be one of the major factors influencing patients' visual quality and satisfaction. The goal of this study is to compare the clinical outcomes of femtosecond laser arcuate keratotomy in one eye and Toric intraocular lens implantation in the contralateral eye for astigmatism correction in patients undergoing femtosecond laser-assisted cataract surgery. The study is a prospective randomized comparative study. Patients with binocular regular corneal astigmatism ranging from 0.75 to 3.00 D will be recruited. The patient will randomly receive femtosecond laser arcuate keratotomy in one eye and receive Toric intraocular lens implantation in the contralateral eye. Long term evaluation will be performed to compare the visual acuity, subjective manifest refraction, and corneal topography between groups.

ELIGIBILITY:
Inclusion Criteria:

* cataract patients
* patients with binocular regular corneal astigmatism ranging from 0.75 to 3.00 D
* patients who plan to receive femtosecond laser-assisted cataract surgery

Exclusion Criteria:

* patients with ocular surface abnormalities such as irregular corneal astigmatism, corneal scarring, keratoconus, and pterygium)
* patients with history of ocular trauma or surgery
* patients with coexisting ocular disorders such as glaucoma, retinal vascular occlusive disease, retinal detachment, diabetic retinopathy, and any optic nerve-related pathologies
* patients with concurrent severe systemic diseases
* patients who lack of cooperation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Refractive astigmatism | 1 day, 1 week, 1 month, 3 months and 1year postoperatively
  subjective manifest refraction and residual astigmatism

SECONDARY OUTCOMES:
Visual acuity | 1 day, 1 week, 1 month, 3 months and 1year postoperatively
  uncorrected distance visual acuity and corrected distance visual acuity

OTHER OUTCOMES:
Keratometric astigmatism | 1 day, 1 week, 1 month, 3 months and 1year postoperatively
  Corneal topography measurement

CONTACTS AND LOCATIONS:
Overall Officials: Ke Yao, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Eye Center of the Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Noh H, Yoo YS, Shin KY, Lim DH, Chung TY. Comparison of penetrating femtosecond laser-assisted astigmatic keratotomy and toric intraocular lens implantation for correction of astigmatism in cataract surgery. Sci Rep. 2021 Apr 1;11(1):7340. doi: 10.1038/s41598-021-86763-5. PMID 33795782
- [Background] Yoo A, Yun S, Kim JY, Kim MJ, Tchah H. Femtosecond Laser-assisted Arcuate Keratotomy Versus Toric IOL Implantation for Correcting Astigmatism. J Refract Surg. 2015 Sep;31(9):574-8. doi: 10.3928/1081597X-20150820-01. PMID 26352561